CLINICAL TRIAL: NCT03019237
Title: The Effect of Intranasal Application of Anti-IgE Antibodies on IgE Production in Patients Suffering From Seasonal Allergic Rhinitis - a Pilot Study
Brief Title: Effect of Intranasal Anti-IgE Antibodies on IgE Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Verena Niederberger-Leppin, ao. Univ.-Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-004193-25
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — anti-IgE antibodies; Omalizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- intranasal anti-IgE (Experimental): Anti-IgE (Xolair) will be freshly diluted in sterile 0.9% sodium chloride solution (438 μg/ml) and will be administered using a metered pump delivering 15 μl per puff to both nostrils on three consecutive days.
  Interventions: Drug: anti-IgE
- intranasal allergen (Active Comparator): GMP produced rBet v 1 will be freshly diluted in sterile 0.9% sodium chloride solution (50 μg/ml) and will be administered using a metered pump delivering 15 μl per puff to both nostrils on three consecutive days.
  Interventions: Other: intranasal allergen
- intranasal saline (Placebo Comparator): Sterile 0.9% sodium chloride solution will be administered using a metered pump delivering 15 μl per puff to both nostrils on three consecutive days.
  Interventions: Other: intranasal saline

INTERVENTIONS:
Drug: anti-IgE — intranasal anti-IgE
  Other Names: Omalizumab
  Arms: intranasal anti-IgE
Other: intranasal allergen — intranasal allergen
  Other Names: GMP produced recombinant Bet v 1
  Arms: intranasal allergen
Other: intranasal saline — intranasal placebo
  Other Names: sodium chloride 0.9%
  Arms: intranasal saline

SUMMARY:
In this study, participants will receive either intranasal anti-IgE-antibodies (n=5) or intranasal allergen (n=5) or intranasal placebo (n=5). Blood samples will be obtained before nasal administration of study drugs and 3, 5 and 8 weeks thereafter. In the serum samples, specific and total IgE levels will be assessed.

DETAILED DESCRIPTION:
The intranasal challenge study will be performed over 8 weeks outside of the birch pollen season (November to January) as a randomized, double blind and placebo-controlled study. During a screening visit, 15 individuals will be recruited according to eligibility criteria. They will be randomized into 3 groups (i.n. administration of anti-IgE antibodies, Bet v 1 or placebo). Intranasal administration will take place on three consecutive days and serum samples will be taken 3, 5, and 8 weeks (+/- 4 days) after the treatment for analysis of total and specific IgE levels

ELIGIBILITY:
Inclusion Criteria:

birch pollen allergy

Exclusion Criteria:

history of anaphylaxis autoimmune diseases treatment with corticosteroids, antihistamines, immunosuppressant drugs, beta-blockers significant medical conditions pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change of allergen-specific IgE | 8 weeks

SECONDARY OUTCOMES:
changes in total IgE | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Verena Niederberger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Otorhinolaryngology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided